CLINICAL TRIAL: NCT07191600
Title: A Study on the Integration of Talking Pen Audio-Interactive Technology With Oral Frailty Delay Care Programs for Enhancing the Physical and Mental Health of Community-Dwelling Elderly: Development, Testing, and Effectiveness Evaluation in Agricultural Counties
Brief Title: Talking Pen Audio-Interactive Program for Oral Frailty Delay in Community-Dwelling Elderly
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113-813
Record Dates: First submitted 2025-08-29; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Oral Health of Older Men
Keywords: Interactive Technology; Community-Dwelling Older Adults; Oral Frailty; Physical Health; Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Participants will receive an oral frailty delay care program integrated with talking pen audio-interactive technology. The program includes bilingual (Mandarin and Taiwanese) teaching materials and structured oral frailty care activities, supported by audio-interactive tools. The intervention is conducted over 3-6 months, with follow-up assessments at baseline, 3 months, and 6 months.
  Interventions: Behavioral: Talking Pen Audio-Interactive Oral Frailty Care Program
- Arm 2 (No Intervention): Participants will continue their usual community activities without exposure to the talking pen audio-interactive oral frailty care program. Assessments will be conducted at baseline, 3 months, and 6 months for comparison with the intervention group.

INTERVENTIONS:
Behavioral: Talking Pen Audio-Interactive Oral Frailty Care Program — Participants in the intervention group will receive a structured oral frailty delay care program integrated with talking pen audio-interactive technology. The program includes bilingual (Mandarin and Taiwanese) teaching materials with audio support to enhance comprehension and engagement. Training sessions will focus on oral frailty prevention, oral function exercises, and related health education. The intervention is delivered over 3 to 6 months, with outcomes measured at baseline, 3 months, and 6 months.
  Arms: Arm 1

SUMMARY:
This study aims to develop and evaluate the effectiveness of a talking pen audio-interactive technology integrated with an oral frailty delay care program for community-dwelling older adults in rural agricultural regions of Chiayi County, Taiwan. The intervention is designed to improve oral function, physical health, and mental well-being. Bilingual (Mandarin and Taiwanese) teaching materials on oral frailty care will be developed. Usability and satisfaction testing will be conducted with older adults at local community bases. A quasi-experimental design will be implemented with 10 participants, who will be randomly assigned to an intervention group or a control group. The intervention group will receive the oral frailty care program with talking pen audio-interactive technology, while the control group will continue with regular community activities. Outcomes, including oral function, physical performance, and mental health, will be measured at baseline, 3 months, and 6 months. This study seeks to provide evidence for innovative, accessible, and sustainable approaches to oral frailty prevention in rural elderly populations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years or older residing in community settings of Chiayi County.
* Able to perform basic self-care.
* No severe swallowing difficulties and not dependent on nasogastric tube feeding.
* Clear consciousness and able to communicate in Mandarin or Taiwanese.
* Willing to provide written informed consent and participate in the study.

Exclusion Criteria:

* Individuals not residing in Chiayi County communities.
* Individuals unable to perform activities of daily living independently or with impaired consciousness.
* Individuals with cognitive impairment or psychiatric disorders that prevent cooperation with study procedures.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Anterior Tongue Pressure | Baseline, 3 months, and 6 months
  Maximum tongue pressure at the anterior tongue will be assessed using the Iowa Oral Performance Instrument (IOPI). Each participant will perform 3 trials with 1-2 minutes rest between trials. The maximum value across 3 trials will be recorded as Pmax.
Change in Posterior Tongue Pressure (Pmax) | Baseline, 3 months, and 6 months.
  Maximum tongue pressure at the posterior tongue will be assessed using the Iowa Oral Performance Instrument (IOPI). Each participant will perform 3 trials with 1-2 minutes rest between trials. The maximum value across 3 trials will be recorded as Pmax.
Change in Lip Muscle Pressure (Pmax) | Baseline, 3 months, and 6 months.
  Maximum tongue pressure at the lip muscles will be assessed using the Iowa Oral Performance Instrument (IOPI). Each participant will perform 3 trials with 1-2 minutes rest between trials. The maximum value across 3 trials will be recorded as Pmax.
Change in Orbicularis Oris Pressure (Pmax) | Baseline, 3 months, and 6 months.
  Maximum tongue pressure at the orbicularis oris will be assessed using the Iowa Oral Performance Instrument (IOPI). Each participant will perform 3 trials with 1-2 minutes rest between trials. The maximum value across 3 trials will be recorded as Pmax.
Change in Oral Moisture | Baseline, 3 months, and 6 months
  Oral moisture will be assessed using a moisture-checking device placed on the tongue surface. Higher values indicate better salivary condition.

IPD SHARING:
Plan to Share IPD: No